CLINICAL TRIAL: NCT06861218
Title: Cerebrospinal Fluid Cytology-guided Intrathecal Chemo-holiday Therapy for EGFR-positive NSCLC Meningeal Metastases: a One-arm, Phase II Clinical Study
Brief Title: Cerebrospinal Fluid Cytology-guided Intrathecal Chemo-holiday Therapy for EGFR-positive NSCLC Leptomeningeal Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Fan Yun, MD, Prof, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH-IRB-2024-1191(IIT)
Record Dates: First submitted 2024-12-30; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Leptomeningeal Metastases
Keywords: Leptomeningeal Metastases; EGFR; Pemetrexed; intrathecal injection; vometinib
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intrathecal injection of pemetrexed and double dose of vometinib (Experimental)
  Interventions: Drug: pemetrexed; Drug: vometinib

INTERVENTIONS:
Drug: pemetrexed — The pemetrexed is administrated by intrathecal injection with a dose of 50mg, once per week for 4 weeks, followed by every four weeks thereafter. The cerebrospinal fluid(CSF) samples are collected every 4 weeks and the cytology examination will be performed. If CSF cytology was negative, CSF cytology was tested again 1 week later. Two negative tests were considered as negative CSF cytology. If the cytology of cerebrospinal fluid was negative after 4 consecutive intrathecal injections, the intrathecal injection should be stopped. If positive, continue to give a intrathecal injection every 4 weeks until CSF cytology is negative. If CSF cytological positivity or worsening of neurological symptoms occurs again during discontinuation, or if new symptoms appear, the intrathecal injection should be resumed every 4 weeks.
Drug: vometinib — double dose of vometinib (160mg)

SUMMARY:
With the rapid development of targeted drugs, the treatment of patients with leptomeningeal metastasis has become a very difficult problem in clinical work. High-dose targeted drugs and intrathecal chemotherapy are important treatment methods for meningeal metastasis. However, it is vital to note that safety is also of concern in previous studies of intrathecal chemotherapy. In this study, we aim to evaluate the safety and effectiveness of patient using chemo-holiday therapy based on the cerebrospinal fluid cytology, combined with double-dose EGFR-targeted drug in patients with leptomeningeal metastases from EGFR-positive NSCLC.

DETAILED DESCRIPTION:
This is a single arm phase II clinical trial. The objective of the study is patients with leptomeningeal metastases from non-small cell lung cancer after EGFR TKIs treatment. The pemetrexed is administrated by intrathecal injection with a dose of 50mg, once per week for 4 weeks, followed by every four weeks thereafter. The cerebrospinal fluid(CSF) samples are collected every 4 weeks and the cytology examination will be performed. If CSF cytology was negative, CSF cytology was tested again 1 week later. Two negative tests were considered as negative CSF cytology. If the cytology of cerebrospinal fluid was negative after 4 consecutive intrathecal injections, the intrathecal injection should be stopped. If positive, continue to give a intrathecal injection every 4 weeks until CSF cytology is negative. If CSF cytological positivity or worsening of neurological symptoms occurs again during discontinuation, or if new symptoms appear, the intrathecal injection should be resumed every 4 weeks. in the meantime, double dose of vometinib (160mg) is given.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18 and 75 years.
2. Histologically or cytologically confirmed diagnosis of NSCLC with EGFR mutations.
3. Cytologically confirmed diagnosis of leptomeningeal metastasis.
4. Normal organ function.
5. No history of severe nervous system disease.
6. No severe dyscrasia.

Exclusion Criteria:

1. Any evidence of nervous system failure, including severe encephalopathy, grade 3 or 4 leukoencephalopathy on imaging, and Glasgow Coma Score less than 11.
2. Any evidence of extensive and lethal progressive systemic diseases without effective treatment.
3. Patients with poor compliance or other reasons that were unsuitable for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the enrollment of this study until date of death from any cause, up to a maximum of approximately 2 years
  Overall survival is the time from the date of enrollment of this study to death due to any cause.

SECONDARY OUTCOMES:
Impact on quality of life | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  Impact on quality of life using QLQ-C30 (V3.0)
Clinical response rate | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The response assessment in neuro-oncology criteria (RANO) proposal for response criteria of leptomeningeal metastasis was used to assess the clinical response in this study.
leptomeningeal metastases related progression-free survival | From date of treatment until the date of first documented neurological progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The neurological progression was determined based on the RANO proposal evaluation criteria which have been established and published on Neuro Oncol.
CSF cytological clearance | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The cerebrospinal fluid samples are collected every 4 weeks and the cytology examination will be performed.
Adverse events | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The incidence of treatment-related adverse events were measured for determining tolerability and safety according to Common Toxicity Criteria Adverse Event (CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China